CLINICAL TRIAL: NCT01285609
Title: Randomized, Multicenter, Double-Blind, Phase 3 Trial Comparing the Efficacy of Ipilimumab in Addition to Paclitaxel and Carboplatin Versus Placebo in Addition to Paclitaxel and Carboplatin in Subjects With Stage IV/Recurrent Non Small Cell Lung Cancer (NSCLC)
Brief Title: Phase 3 Trial in Squamous Non Small Cell Lung Cancer Subjects Comparing Ipilimumab Versus Placebo in Addition to Paclitaxel and Carboplatin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA184-104; 2009-017396-19 (EudraCT Number)
Record Dates: First submitted 2011-01-24; First posted 2011-01-28 (Estimated); Results first posted 2016-06-23 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Lung Cancer - Non Small Cell Squamous
MeSH Terms: interventions — Ipilimumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ipilimumab + Paclitaxel and Carboplatin (Experimental): Ipilimumab + Active Chemo Backbone
  Ipilimumab: IV solution, intravenous (IV), 10 mg/kg, 90 minute infusion, Once every 3 weeks for 4 doses and then every 12 weeks until disease progression (for a maximum treatment period of 3 years from the first dose)
  Paclitaxel: IV solution, IV, 175 mg/m², 3 hour infusion, Once every 3 weeks for 6 doses
  Carboplatin: IV solution, IV, Area Under the Curve (AUC) = 6, 30 minute infusion, Once every 3 weeks for 6 doses
  Interventions: Drug: Ipilimumab; Drug: Paclitaxel; Drug: Carboplatin
- Placebo + Paclitaxel and Carboplatin (Placebo Comparator): Placebo + Active Chemo Backbone
  Placebo: IV solution, IV, 0.9% sodium chloride or 5% dextrose, 90 minute infusion, Once every 3 weeks for 4 doses and then every 12 weeks until disease progression (for a maximum treatment period of 3 years from the first dose)
  Paclitaxel: IV solution, IV, 175 mg/m², 3 hour infusion, Once every 3 weeks for 6 doses
  Carboplatin: IV solution, IV, Area Under the Curve (AUC) = 6, 30 minute infusion, Once every 3 weeks for 6 doses
  Interventions: Drug: Placebo; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Ipilimumab
  Other Names: BMS-734016
  Arms: Ipilimumab + Paclitaxel and Carboplatin
Drug: Placebo
  Arms: Placebo + Paclitaxel and Carboplatin
Drug: Paclitaxel
  Other Names: Taxol®
Drug: Carboplatin
  Other Names: Paraplatin®

SUMMARY:
The purpose of the study is to determine whether Ipilimumab plus Paclitaxel and Carboplatin will extend the lives of patients with squamous only non small cell lung cancer more than placebo plus Paclitaxel and Carboplatin.

DETAILED DESCRIPTION:
The primary objective is to compare Overall Survival (OS) of participants with Stage IV/recurrent NSCLC of squamous histology who have been randomized to ipilimumab in addition to paclitaxel and carboplatin versus placebo in addition to paclitaxel and carboplatin, and have received at least one dose of blinded study therapy (ipilimumab or placebo).

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Non small cell lung cancer (NSCLC) - squamous cell
* Stage IV or recurrent NSCLC
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Brain Metastases
* Autoimmune diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1289 (Actual)
Dates: Start 2011-01-16 (Actual); Primary Completion 2015-06-09 (Actual); Study Completion 2017-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (251):
- United States (33):
  - Sharp Memorial Hospital, San Diego, California
  - Va Connecticut Healthcare System, West Haven, Connecticut
  - Lynn Cancer Institute Center For Hematology-Oncology, Boca Raton, Florida
  - Integrated Community Oncology Network, Jacksonville, Florida
  - University Of Illinois At Chicago Medical Center, Chicago, Illinois
  - Quincy Medical Group, Quincy, Illinois
  - Presence Medical Group Hematology Oncology, Skokie, Illinois
  - Southern Illinois University School Of Medicine, Springfield, Illinois
  - St. Francis Hospital & Health Centers, Indianapolis, Indiana
  - Floyd Memorial Cancer Center Of Indiana, New Albany, Indiana
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Montgomery Cancer Center, Mount Sterling, Kentucky
  - St Joseph Mercy Hospital, Ypsilanti, Michigan
  - University Of Kansas Cancer Center, Kansas City, Missouri
  - Washington University School Of Medicine, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Clinical Research Alliance, Inc., Lake Success, New York
  - Durham Va Medical Center (111g), Durham, North Carolina
  - Carolina Biooncology Institute, Huntersville, North Carolina
  - Novant Health Oncology Specialists, Lexington, North Carolina
  - Gabrail Cancer Center Research, Canton, Ohio
  - Oklahoma Oncology And Hematology, Pc Dba, Tulsa, Oklahoma
  - Kaiser Permanente Northwest Region, Portland, Oregon
  - Guthrie Medical Group, P.C., Sayre, Pennsylvania
  - Wjb Dorn Va Medical Center, Columbia, South Carolina
  - Cancer Center Of The Carolinas, Greenville, South Carolina
  - Associated in Oncology and Hematology, Chattanooga, Tennessee
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - Thompson Oncology Group, Knoxville, Tennessee
  - Texas Oncology, PA - South Austin Cancer Center, Austin, Texas
  - Blue Ridge Cancer Care, Blacksburg, Virginia
  - Wisconsin Institutes for Medical Research, Madison, Wisconsin
- Argentina (6):
  - Local Institution, Quilmes, Buenos Aires
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, San Miguel de Tucumán, Tucumán Province
  - Local Institution, Córdoba
  - Local Institution, Mendoza
  - Local Institution, Santa Fe
- Australia (5):
  - Local Institution, Bedford Park, South Australia
  - Local Institution, Box Hill, Victoria
  - Local Institution, Frankston, Victoria
  - Local Institution, Heidelberg, Victoria
  - Local Institution, Wodonga, Victoria
- Austria (3):
  - Local Institution, Graz
  - Local Institution, Linz
  - Local Institution, Salzburg
- Belgium (4):
  - Local Institution, Aalst
  - Local Institution, Liège
  - Local Institution, Sint-Niklaas
  - Local Institution, Yvoir
- Brazil (10):
  - Local Institution, Fortaleza, Ceará
  - Local Institution, Belo Horizonte, Minas Gerais
  - Local Institution, Curitiba, Paraná
  - Local Institution, Passo Fundo, Rio Grande do Sul
  - Local Institution, Barretos, São Paulo
  - Local Institution, São José dos Campos, São Paulo
  - Local Institution, Porto Alegre
  - Local Institution, Ribeirão Preto
  - Local Institution, Rio de Janeiro
  - Local Institution, São Paulo
- Canada (2):
  - Local Institution, Montreal, Quebec
  - Local Institution, Oshawa
- Chile (2):
  - Local Institution, Viña del Mar, Región de Valparaíso
  - Local Institution, Santiago, Santiago Metropolitan
- China (13):
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Guanzhou, Guangdong
  - Local Institution, Shantou, Guangdong
  - Local Institution, Wuhan, Hubei
  - Local Institution, Nanjing, Jiangsu
  - Local Institution, Suzhou, Jiangsu
  - Local Institution, Changchun, Jilin
  - Local Institution, Xi'an, Shaanxi
  - Local Institution, Ürümqi, Xinjiang
  - Local Institution, Hangzhou, Zhejiang
  - Local Institution, Beijing
  - Local Institution, Santiago
  - Local Institution, Shanghai
- Colombia (2):
  - Local Institution, Montería, Departamento de Córdoba
  - Local Institution, Pereira, Risaralda Department
- Czechia (5):
  - Local Institution, Ostrava, Poruba
  - Local Institution, Prague
  - Local Institution, Pribram V-Zdabor
  - Local Institution, Ústí nad Labem
  - Local Institution, Znojmo
- Denmark (5):
  - Local Institution, Aalborg
  - Local Institution, Herlev
  - Local Institution, Hillerød
  - Local Institution, Næstved
  - Local Institution, Odense
- France (7):
  - Local Institution, Caen
  - Local Institution, Marseille
  - Local Institution, Paris
  - Local Institution, Poitiers
  - Local Institution, Rennes
  - Local Institution, Toulouse
  - Local Institution, Vandœuvre-lès-Nancy
- Germany (19):
  - Local Institution, Bad Berka
  - Local Institution, Bochum
  - Local Institution, Darmstadt
  - Local Institution, Dresden
  - Local Institution, Frankfurt am Main
  - Local Institution, Gauting
  - Local Institution, Grosshandsdorf
  - Local Institution, Hamburg
  - Local Institution, Heidelberg
  - Local Institution, Kassel
  - Local Institution, Lübeck
  - Local Institution, Mainz
  - Local Institution, München
  - Local Institution, Neumünster
  - Local Institution, Nuremberg
  - Local Institution, Regensburg
  - Local Institution, Tübingen
  - Local Institution, Ulm
  - Local Institution, Villingen-Schwenningen
- Hong Kong (2):
  - Local Institution, Hong Kong
  - Local Institution, New Territories
- Hungary (10):
  - Local Institution, Budapest
  - Local Institution, Deszk
  - Local Institution, Farkasgyepű
  - Local Institution, Gyula
  - Local Institution, Mátraháza
  - Local Institution, Nyíregyháza
  - Local Institution, Pécs
  - Local Institution, Sopron
  - Local Institution, Székesfehérvár
  - Local Institution, Szolnok
- Ireland (2):
  - Local Institution, Dublin
  - Local Institution, Galway
- Israel (9):
  - Local Institution, Beersheba
  - Local Institution, Haifa
  - Local Institution, Jerusalem
  - Local Institution, Nahariya
  - Local Institution, Petah Tikva
  - Local Institution, Rehovot
  - Local Institution, Tel Aviv
  - Local Institution, Tel Litwinsky
  - Local Institution, Ẕerifin
- Italy (11):
  - Local Institution, Benevento
  - Local Institution, Bologna
  - Local Institution, Lido di Camaiore
  - Local Institution, Lucca
  - Local Institution, Monza
  - Local Institution, Padua
  - Local Institution, Perugia
  - Local Institution, Siena
  - Local Institution, Sondrio
  - Local Institution, Terni
  - Local Institution, Treviglio
- Japan (20):
  - Local Institution, Nagoya, Aichi-ken
  - Local Institution, Kashiwa, Chiba
  - Local Institution, Kanazawa, Ishikawa-ken
  - Local Institution, Yokohama, Kanagawa
  - Local Institution, Natori-shi, Miyagi
  - Local Institution, Sendai, Miyagi
  - Local Institution, Kurashiki-shi, Okayama-ken
  - Local Institution, Hirakata-shi, Osaka
  - Local Institution, Osaka, Osaka
  - Local Institution, Sunto-gun, Shizuoka
  - Local Institution, Chuo-ku, Tokyo
  - Local Institution, Ube-shi, Yamaguchi
  - Local Institution, Akashi, Hyogo
  - Local Institution, Fukuoka
  - Local Institution, Matsuyama, Ehime
  - Local Institution, Sapporo Hokkaido
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Sayama
  - Local Institution, Takatsuki
  - Local Institution, Tokyo
- Mexico (3):
  - Local Institution, Zapopan, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Monterrey, Nuevo León
- Netherlands (4):
  - Local Institution, 's-Hertogenbosch
  - Local Institution, Breda
  - Local Institution, Harderwijk
  - Local Institution, Nieuwegein
- Peru (4):
  - Local Institution, Trujillo, La Libertad
  - Local Institution, Arequipa
  - Local Institution, Cercado
  - Local Institution, Lima
- Poland (10):
  - Local Institution, Elblag
  - Local Institution, Gdansk
  - Local Institution, Gdansk- Zaspa
  - Local Institution, Grudziądz
  - Local Institution, Olsztyn
  - Local Institution, Otwock
  - Local Institution, Poznan
  - Local Institution, Szczecin
  - Local Institution, Torun
  - Local Institution, Warsaw
- Portugal (5):
  - Local Institution, São Martinho do Bispo, Coimbra District
  - Local Institution, Lisbon
  - Local Institution, Porto
  - Local Institution, Santa Maria da Feira
  - Local Institution, Vila Nova de Gaia
- Romania (5):
  - Local Institution, Bucharest
  - Local Institution, Cluj-Napoca
  - Local Institution, Sibiu
  - Local Institution, Suceava
  - Local Institution, Timișoara
- Russia (7):
  - Local Institution, Chelyabinsk
  - Local Institution, Kazan'
  - Local Institution, Moscow
  - Local Institution, Pyatigorsk
  - Local Institution, Saint Petersburg
  - Local Institution, St-Peterburg
  - Local Institution, Tula
- Local Institution, Singapore, Singapore
- South Africa (4):
  - Local Institution, Vereeniging, Gauteng
  - Local Institution, Panorama,cape Town, Western Cape
  - Local Institution, Cape Town
  - Local Institution, Durban
- South Korea (10):
  - Local Institution, Goyang-si, Gyeonggi-do
  - Local Institution, Suwon, Gyeonggi-do
  - Local Institution, Seoul, Kangnam-gu
  - Local Institution, Cheonju-si, North Chungcheong
  - Local Institution, Seoul, Seodaemungu
  - Local Institution, Busan
  - Local Institution, Daegu
  - Local Institution, Gyeonggi-do
  - Local Institution, Seoul
  - Local Institution, Suwon
- Spain (8):
  - Local Institution, Barakaldo, Vizcaya
  - Local Institution, Ávila
  - Local Institution, Benidorm-alicante
  - Local Institution, Castellon
  - Local Institution, Madrid
  - Local Institution, Manresa
  - Local Institution, Ourense
  - Local Institution, Valencia
- Sweden (4):
  - Local Institution, Gothenburg
  - Local Institution, Lund
  - Local Institution, Stockholm
  - Local Institution, Umeå
- Switzerland (2):
  - Local Institution, Basel
  - Local Institution, Winterthur
- Taiwan (5):
  - Local Institution, Changhua
  - Local Institution, Chiayi City
  - Local Institution, Kaohsiung County
  - Local Institution, Taichung
  - Local Institution, Taipei
- Thailand (4):
  - Local Institution, Bangkok, Tungpayathai
  - Local Institution, Bangkok
  - Local Institution, Chiang Mai
  - Local Institution, Songkhla
- United Kingdom (5):
  - Local Institution, Dundee, Angus/forfarshire
  - Local Institution, Truro, Cornwall
  - Local Institution, Southampton, Hampshire
  - Local Institution, Nottingham
  - Local Institution, Sheffield

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1289 participants were enrolled and 956 were randomized (479 Ipilimumab, 477 Placebo). 948 were treated (475 Ipilimumab, 473 Placebo). Reasons for non-treatment is 4 no longer met study criteria, 2 adverse events unrelated to study drug, 1 participant request to discontinue, and 1 other.
Groups:
- Ipilimumab With Paclitaxel/Carboplatin: Ipilimumab + Active Chemotherapy Backbone The blinded therapy (Ipilimumab) started at the 3rd dose of active chemotherapy backbone (Paclitaxel/Carboplatin). Ipilimumab: IV solution, intravenous (IV), 10 mg/kg, 90 minute infusion, Once every 3 weeks for 4 doses and then every 12 weeks until disease progression (for a maximum treatment period of 3 years from the first dose) Active Chemo Backbone: Paclitaxel: IV solution, IV, 175 mg/m², 3 hour infusion, Once every 3 weeks for 6 doses Carboplatin: IV solution, IV, Area Under the Curve (AUC) = 6, 30 minute infusion, Once every 3 weeks for 6 doses
- Placebo With Paclitaxel/Carboplatin: Placebo + Active Chemotherapy Backbone The blinded therapy (Placebo) started at the 3rd dose of active chemotherapy backbone (Paclitaxel/Carboplatin). Placebo: IV solution, IV, 0.9% sodium chloride or 5% dextrose, 90 minute infusion, Once every 3 weeks for 4 doses and then every 12 weeks until disease progression (for a maximum treatment period of 3 years from the first dose) Active Chemotherapy Backbone: Paclitaxel: IV solution, IV, 175 mg/m², 3 hour infusion, Once every 3 weeks for 6 doses Carboplatin: IV solution, IV, Area Under the Curve (AUC) = 6, 30 minute infusion, Once every 3 weeks for 6 doses
Period: Randomized
Arm/Group | Ipilimumab With Paclitaxel/Carboplatin | Placebo With Paclitaxel/Carboplatin
Started (Started = Randomized) | 479 (Represents participants randomized to this arm prior to 1st dose of chemotherapy treatment) | 477 (Represents participants randomized to this arm prior to 1st dose of chemotherapy treatment)
Treated With Chemotherapy (1st Dose) | 475 | 473
Completed (Completed = Continued to Blinded Therapy) | 388 | 361
Not Completed | 91 | 116
Not completed — Progressive Disease | 41 | 61
Not completed — Adverse Event Unrelated to Study Drug | 18 | 18
Not completed — Study Drug Toxicity | 13 | 14
Not completed — Death | 5 | 7
Not completed — Withdrawal by Subject | 8 | 11
Not completed — Subject No Longer Met Study Criteria | 1 | 1
Not completed — Undisclosed Reasons | 1 | 0
Not completed — Randomized but not Treated | 4 | 4
Period: Treated With Blinded Therapy
Arm/Group | Ipilimumab With Paclitaxel/Carboplatin | Placebo With Paclitaxel/Carboplatin
Started (Started = Received at least one dose of Blinded Therapy) | 388 | 361
Completed (Completed = Completed the Blinded Therapy treatment phase) | 1 | 2
Not Completed | 387 | 359
Not completed — Progressive Disease | 223 | 305
Not completed — Study Drug Toxicity | 87 | 14
Not completed — Adverse Event Unrelated to Study Drug | 36 | 14
Not completed — Withdrawal by Subject | 20 | 7
Not completed — Death | 11 | 3
Not completed — Maximum Clinical Benefit | 2 | 4
Not completed — Not Reported | 0 | 2
Not completed — Poor/Non-Compliance | 1 | 2
Not completed — Subject No Longer Met Study Criteria | 1 | 0
Not completed — Administrative Reason by Sponsor | 1 | 3
Not completed — Physician and Patient decision | 1 | 3
Not completed — Participant refused participation | 1 | 0
Not completed — Participant started radiotherapy | 1 | 0
Not completed — Participant hospitalized | 1 | 0
Not completed — Investigator's assessment | 1 | 0
Not completed — PI decision to discontinue | 0 | 1
Not completed — Worsening of general condition | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized Participants Who Received at Least One Dose of Blinded Study Therapy
Groups:
- Ipilimumab With Paclitaxel/Carboplatin: Ipilimumab + Active Chemo Backbone The blinded therapy (Ipilimumab) started at the 3rd dose of active chemotherapy backbone (Paclitaxel/Carboplatin). Ipilimumab: IV solution, intravenous (IV), 10 mg/kg, 90 minute infusion, Once every 3 weeks for 4 doses and then every 12 weeks until disease progression (for a maximum treatment period of 3 years from the first dose) Active Chemo Backbone: Paclitaxel: IV solution, IV, 175 mg/m², 3 hour infusion, Once every 3 weeks for 6 doses Carboplatin: IV solution, IV, Area Under the Curve (AUC) = 6, 30 minute infusion, Once every 3 weeks for 6 doses
- Placebo With Paclitaxel/Carboplatin: Placebo + Active Chemo Backbone The blinded therapy (Placebo) started at the 3rd dose of active chemotherapy backbone (Paclitaxel/Carboplatin). Placebo: IV solution, IV, 0.9% sodium chloride or 5% dextrose, 90 minute infusion, Once every 3 weeks for 4 doses and then every 12 weeks until disease progression (for a maximum treatment period of 3 years from the first dose) Active Chemo Backbone: Paclitaxel: IV solution, IV, 175 mg/m², 3 hour infusion, Once every 3 weeks for 6 doses Carboplatin: IV solution, IV, Area Under the Curve (AUC) = 6, 30 minute infusion, Once every 3 weeks for 6 doses
- Total: Total of all reporting groups
Arm/Group | Ipilimumab With Paclitaxel/Carboplatin | Placebo With Paclitaxel/Carboplatin | Total
Number analyzed (Participants) | 388 | 361 | 749
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (8.27) | 63.7 (8.70) | 63.7 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 52 | 114
  Male | 326 | 309 | 635
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 106 | 108 | 214
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 276 | 243 | 519
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 6 | 9
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG Performance Status is a 6-item scale used to assess disease progression, daily functioning, appropriate treatment, and prognosis. Performance status is scored on a scale ranging from 0-5, with (best score) 0=fully active and able to carry on all pre-disease performance without restriction and (worst score) 5=death.
  Participants
    0 | 135 | 124 | 259
    1 | 251 | 234 | 485
    2 | 1 | 3 | 4
    3 | 1 | 0 | 1
Disease Stage at Study Entry [Count of Participants; unit: Participants] — Non-Small Cell Lung Cancer is categorized in 4 Stages (I-IV). I: Cancer located only in lungs and has not spread to any lymph nodes. II: Cancer in the lung and nearby lymph nodes. III: Cancer in the lung and lymph nodes in the middle of the chest. Stage III has two subtypes, IIIA (cancer has spread only to lymph nodes on the same side of the chest where the cancer started) and IIIB (cancer has spread to the lymph nodes on the opposite side of the chest, or above the collar bone). IV: Cancer has spread to both lungs, to fluid in the area around the lungs, or to another part of the body.
  Participants
    Stage IV | 367 | 333 | 700
    Recurrent | 21 | 28 | 49

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) in Participants Who Received at Least One Dose of Blinded Study Therapy at Primary Endpoint
Description: Overall Survival (OS) was defined as the time from randomization to the date of death. Participants that had not died were censored at last known date alive. Median OS time was calculated using Kaplan-Meier Estimates. Analysis for the Primary Endpoint occurred when the following 2 conditions were both met: (1) 518 deaths were observed in randomized participants treated with at least one dose of blinded study therapy and (2) 705 deaths were observed in all randomized participants.
Time Frame: Randomization until 518 deaths were observed in randomized participants treated with at least one dose of blinded study therapy and 705 deaths were observed in all randomized participants, up to June 2015 (approximately 48 months post study start)
Population: All treated participants who received at least one dose of blinded therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab With Paclitaxel/Carboplatin | Placebo With Paclitaxel/Carboplatin
Number analyzed (Participants) | 388 | 361
months | 13.37 [11.76 to 14.78] | 12.42 [11.60 to 13.63]
Statistical Analysis 1: Comparison: Ipilimumab With Paclitaxel/Carboplatin vs Placebo With Paclitaxel/Carboplatin; Hazard ratio = Ipilimumab with Paclitaxel/Carboplatin over Placebo with Paclitaxel/Carboplatin; Test type: Superiority or Other; p = 0.2517, Log Rank; p-value based on an unstratified 2-sided log rank test; Hazard Ratio (HR) = 0.907, 95% CI 2-sided [0.767 to 1.072] — Hazard of Ipilimumab over Hazard of Placebo with 2-sided 95% confidence intervals are based on an unstratified Cox proportional hazards model with treatment as the single covariate

2. Secondary Outcome: Overall Survival (OS) in All Randomized Participants at Primary Endpoint
Description: as for outcome 1
Time Frame: as for outcome 1
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipilimumab With Paclitaxel/Carboplatin | Placebo With Paclitaxel/Carboplatin
Number analyzed (Participants) | 479 | 477
months | 10.94 [9.56 to 12.02] | 10.74 [9.66 to 11.73]
Statistical Analysis 1: Comparison: Ipilimumab With Paclitaxel/Carboplatin vs Placebo With Paclitaxel/Carboplatin; Hazard ratio = Ipilimumab with Paclitaxel/Carboplatin over Placebo with Paclitaxel/Carboplatin; Test type: Superiority or Other; p = 0.2421, Log Rank — p-value based on stratified 2-sided log-rank test; Hazard Ratio (HR) = 0.917, 95% CI 2-sided [0.792 to 1.061] — Hazard of Ipilimumab over Placebo with 2-sided 95% confidence intervals based on a stratified Cox proportional hazards model with several stratification factors and treatment as the single covariate

3. Secondary Outcome: Median Number of Months With Progression Free Survival (PFS) Per mWHO in Participants Who Have Received at Least One Dose of Blinded Study Therapy at Primary Endpoint
Description: Progression-free survival (PFS) is defined as the time between the date of randomization and the date of tumor progression per Modified World Health Organization (mWHO) criteria or death, whichever occurs first. A participant who died without reported progression per mWHO criteria were considered to have progressed on the date of death. For participants who remain alive and have not progressed, PFS was censored on the date of last evaluable tumor assessment. For participants who remain alive and have no recorded post-baseline tumor assessment, PFS was censored on the day of randomization.
Time Frame: as for outcome 1
Population: All treated participants who received at least one dose of blinded therapy
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Ipilimumab With Paclitaxel/Carboplatin: Ipilimumab + Active Chemo Backbone The blinded therapy (Ipilimumab) started at the 3rd dose of active chemotherapy backbone (Paclitaxel/Carboplatin). Ipilimumab: IV solution, intravenous (IV), 10 mg/kg, 90 minute infusion, Once every 3 weeks for 4 doses and then every 12 weeks until disease progression (for a maximum treatment period of 3 years from the first dose) Active Chemotherapy Backbone: Paclitaxel: IV solution, IV, 175 mg/m², 3 hour infusion, Once every 3 weeks for 6 doses Carboplatin: IV solution, IV, Area Under the Curve (AUC) = 6, 30 minute infusion, Once every 3 weeks for 6 doses
- Placebo With Paclitaxel/Carboplatin: Placebo + Active Chemo Backbone The blinded therapy (Placebo) started at the 3rd dose of active chemotherapy backbone (Paclitaxel/Carboplatin). Placebo: IV solution, IV, 0.9% sodium chloride or 5% dextrose, 90 minute infusion, Once every 3 weeks for 4 doses and then every 12 weeks until disease progression (for a maximum treatment period of 3 years from the first dose) Active Chemotherapy Backbone: Paclitaxel: IV solution, IV, 175 mg/m², 3 hour infusion, Once every 3 weeks for 6 doses Carboplatin: IV solution, IV, Area Under the Curve (AUC) = 6, 30 minute infusion, Once every 3 weeks for 6 doses
Arm/Group | Ipilimumab With Paclitaxel/Carboplatin | Placebo With Paclitaxel/Carboplatin
Number analyzed (Participants) | 388 | 361
months | 5.55 [5.36 to 5.85] | 5.59 [5.52 to 5.72]
Statistical Analysis 1: Comparison: Ipilimumab With Paclitaxel/Carboplatin vs Placebo With Paclitaxel/Carboplatin; Hazard ratio = Ipilimumab with Paclitaxel/Carboplatin over Placebo with Paclitaxel/Carboplatin; Test type: Superiority or Other; p = 0.0678, Log Rank; p-value based on an unstratified 2-sided log rank test; Hazard Ratio (HR) = 0.869, 95% CI 2-sided [0.749 to 1.009] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Day of first dose to 90 days post final dose, up to August 2017 (approximately 72 months post study start)
Groups:
- 10 MG/KG Ipilimumab + Paclitaxel/ Carbop: Ipilimumab + Active Chemotherapy Backbone The blinded therapy (Ipilimumab) started at the 3rd dose of active chemotherapy backbone (Paclitaxel/Carboplatin). Ipilimumab: IV solution, intravenous (IV), 10 mg/kg, 90 minute infusion, Once every 3 weeks for 4 doses and then every 12 weeks until disease progression (for a maximum treatment period of 3 years from the first dose) Active Chemo Backbone: Paclitaxel: IV solution, IV, 175 mg/m², 3 hour infusion, Once every 3 weeks for 6 doses Carboplatin: IV solution, IV, Area Under the Curve (AUC) = 6, 30 minute infusion, Once every 3 weeks for 6 doses
- Placebo + Paclitaxel/ Carboplatin: Placebo + Active Chemotherapy Backbone The blinded therapy (Placebo) started at the 3rd dose of active chemotherapy backbone (Paclitaxel/Carboplatin). Placebo: IV solution, IV, 0.9% sodium chloride or 5% dextrose, 90 minute infusion, Once every 3 weeks for 4 doses and then every 12 weeks until disease progression (for a maximum treatment period of 3 years from the first dose) Active Chemotherapy Backbone: Paclitaxel: IV solution, IV, 175 mg/m², 3 hour infusion, Once every 3 weeks for 6 doses Carboplatin: IV solution, IV, Area Under the Curve (AUC) = 6, 30 minute infusion, Once every 3 weeks for 6 doses
Arm/Group | 10 MG/KG Ipilimumab + Paclitaxel/ Carbop | Placebo + Paclitaxel/ Carboplatin
All-Cause Mortality (participants affected / at risk) | 359/475 | 371/473
Serious Adverse Events (participants affected / at risk) | 300/475 | 235/473
Other Adverse Events (participants affected / at risk) | 437/475 | 428/473
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 10 MG/KG Ipilimumab + Paclitaxel/ Carbop (N=475) | Placebo + Paclitaxel/ Carboplatin (N=473)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 21 | 10
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Autoimmune colitis (Gastrointestinal disorders) | 2 | 1
Blood pressure decreased (Investigations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 2
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Completed suicide (Psychiatric disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Device related infection (Infections and infestations) | 1 | 1
Haemoglobin decreased (Investigations) | 1 | 2
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Overdose (Injury, poisoning and procedural complications) | 1 | 5
Performance status decreased (General disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Spinal cord paralysis (Nervous system disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Asbestosis (Injury, poisoning and procedural complications) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Asthenia (General disorders) | 5 | 7
Atrial flutter (Cardiac disorders) | 1 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Blood creatinine increased (Investigations) | 5 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Chest pain (General disorders) | 1 | 4
Cholestasis (Hepatobiliary disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 14 | 2
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Device dislocation (General disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0
Embolism venous (Vascular disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
General physical health deterioration (General disorders) | 7 | 10
Haematemesis (Gastrointestinal disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 3 | 1
Liver disorder (Hepatobiliary disorders) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 35 | 37
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 3
Peripheral ischaemia (Vascular disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pupils unequal (Eye disorders) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 1 | 1
Swelling (General disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Weight decreased (Investigations) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 5 | 8
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 3
Cardio-respiratory arrest (Cardiac disorders) | 5 | 2
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Disease progression (General disorders) | 4 | 5
Fulminant type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Hydrocholecystis (Hepatobiliary disorders) | 0 | 1
Hypertension (Vascular disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophysitis (Endocrine disorders) | 2 | 0
Ileal perforation (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 5
Nasopharyngitis (Infections and infestations) | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Peripheral embolism (Vascular disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 11 | 10
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 11
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Viraemia (Infections and infestations) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Adrenocortical insufficiency acute (Endocrine disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Death (General disorders) | 10 | 7
Drug hypersensitivity (Immune system disorders) | 3 | 1
Empyema (Infections and infestations) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Extravasation (General disorders) | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 9 | 10
Heart injury (Injury, poisoning and procedural complications) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 2
Infection (Infections and infestations) | 3 | 4
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lung squamous cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 2
Platelet count decreased (Investigations) | 1 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pyrexia (General disorders) | 21 | 14
Red blood cell count decreased (Investigations) | 0 | 1
Renal failure (Renal and urinary disorders) | 4 | 2
Septic shock (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 6 | 5
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Body temperature increased (Investigations) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 2
Cholangitis (Hepatobiliary disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 8 | 7
Depression (Psychiatric disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 17 | 16
Embolism (Vascular disorders) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Hypopituitarism (Endocrine disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 3
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 3 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Lung abscess (Infections and infestations) | 3 | 1
Lung infection (Infections and infestations) | 9 | 5
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 8
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Orchitis (Infections and infestations) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Perivascular dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Thyroiditis (Endocrine disorders) | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Adrenal insufficiency (Endocrine disorders) | 2 | 0
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 1
Brain injury (Nervous system disorders) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 2 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 1
Chills (General disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Delirium (Psychiatric disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 2
Gastroenteritis (Infections and infestations) | 1 | 2
Hypersomnia (Nervous system disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Laryngitis (Infections and infestations) | 0 | 1
Liver function test abnormal (Investigations) | 3 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Nephropathy (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 0 | 1
Pain (General disorders) | 3 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Pneumococcal infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 37 | 34
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Rash (Skin and subcutaneous tissue disorders) | 6 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 4
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Syncope (Nervous system disorders) | 3 | 1
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Vena cava thrombosis (Vascular disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0
Brain herniation (Injury, poisoning and procedural complications) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiac arrest (Cardiac disorders) | 2 | 2
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 2
Device occlusion (General disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 37 | 10
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0
Fatigue (General disorders) | 8 | 7
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypothalamo-pituitary disorder (Endocrine disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Renal function test abnormal (Investigations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 2
Sepsis (Infections and infestations) | 7 | 7
Spinal column injury (Injury, poisoning and procedural complications) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Sudden death (General disorders) | 3 | 1
Superior vena cava occlusion (Vascular disorders) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Tumour perforation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 3 | 2
Blood glucose increased (Investigations) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 3 | 4
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1
Endocrine disorder (Endocrine disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Facial paresis (Nervous system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 20 | 11
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
General physical condition abnormal (Investigations) | 2 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 2
Ileus (Gastrointestinal disorders) | 0 | 3
Infectious colitis (Infections and infestations) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multi-organ failure (General disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 16 | 9
Neutropenic sepsis (Infections and infestations) | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1
Pharyngitis (Infections and infestations) | 2 | 0
Phlebitis superficial (Vascular disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 1 | 1
Pulmonary artery stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 2
Seizure (Nervous system disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Ulcerative keratitis (Eye disorders) | 1 | 0
Guillain-barre syndrome (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 10 MG/KG Ipilimumab + Paclitaxel/ Carbop (N=475) | Placebo + Paclitaxel/ Carboplatin (N=473)
Anaemia (Blood and lymphatic system disorders) | 171 | 157
Decreased appetite (Metabolism and nutrition disorders) | 145 | 116
Haemoglobin decreased (Investigations) | 38 | 30
Myalgia (Musculoskeletal and connective tissue disorders) | 66 | 61
Oedema peripheral (General disorders) | 25 | 31
Peripheral sensory neuropathy (Nervous system disorders) | 71 | 98
White blood cell count decreased (Investigations) | 25 | 31
Aspartate aminotransferase increased (Investigations) | 34 | 20
Asthenia (General disorders) | 80 | 55
Bone pain (Musculoskeletal and connective tissue disorders) | 32 | 26
Chest pain (General disorders) | 26 | 45
Paraesthesia (Nervous system disorders) | 20 | 28
Weight decreased (Investigations) | 44 | 27
Headache (Nervous system disorders) | 30 | 22
Leukopenia (Blood and lymphatic system disorders) | 44 | 54
Thrombocytopenia (Blood and lymphatic system disorders) | 77 | 70
Alopecia (Skin and subcutaneous tissue disorders) | 181 | 175
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 34 | 41
Hypomagnesaemia (Metabolism and nutrition disorders) | 27 | 15
Insomnia (Psychiatric disorders) | 61 | 49
Mucosal inflammation (General disorders) | 10 | 27
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 20 | 24
Neuropathy peripheral (Nervous system disorders) | 61 | 57
Platelet count decreased (Investigations) | 47 | 32
Pyrexia (General disorders) | 91 | 70
Vomiting (Gastrointestinal disorders) | 89 | 68
Abdominal pain upper (Gastrointestinal disorders) | 24 | 23
Alanine aminotransferase increased (Investigations) | 37 | 26
Dehydration (Metabolism and nutrition disorders) | 24 | 7
Dizziness (Nervous system disorders) | 35 | 58
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 94 | 97
Hyponatraemia (Metabolism and nutrition disorders) | 37 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 78 | 27
Arthralgia (Musculoskeletal and connective tissue disorders) | 77 | 58
Cough (Respiratory, thoracic and mediastinal disorders) | 82 | 85
Hypokalaemia (Metabolism and nutrition disorders) | 51 | 31
Rash (Skin and subcutaneous tissue disorders) | 87 | 45
Back pain (Musculoskeletal and connective tissue disorders) | 34 | 38
Constipation (Gastrointestinal disorders) | 117 | 103
Diarrhoea (Gastrointestinal disorders) | 145 | 89
Fatigue (General disorders) | 142 | 140
Abdominal pain (Gastrointestinal disorders) | 25 | 26
Nausea (Gastrointestinal disorders) | 152 | 151
Neutropenia (Blood and lymphatic system disorders) | 107 | 102
Neutrophil count decreased (Investigations) | 31 | 31
Pain in extremity (Musculoskeletal and connective tissue disorders) | 43 | 43
Stomatitis (Gastrointestinal disorders) | 27 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.